CLINICAL TRIAL: NCT04537364
Title: Protocol for a Cohort Diagnostic Accuracy Study to Develop Prediction of Renal Parenchymal Damage and to Evaluate Accuracy of Renal Function in Congenital Anomalies of the Kidney and Urinary Tract (CAKUT)
Brief Title: Prediction of Renal Parenchymal Damage of CAKUT
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: RPD-CAKUT1
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: CAKUT
MeSH Terms: conditions — Cakut

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pediatric patients with CAKUT: This cohort is composed of pediatric children diagnosed of CAKUT from Shanghai peri-conceptional parent-offspring cohort (SPCC) clinic research related outpatient and high-risk newborns referral outpatient, and those who are enrolled in nephrology department and urinary surgery department with CAKUT diagnosis.
  By diagnostic tests for predicting renal parenchymal damage in this cohort, data of kidney images, urinary biomarkers and disease genes can be collected.
  Interventions: Diagnostic Test: combined diagnosis of renal parenchymal damage

INTERVENTIONS:
Diagnostic Test: combined diagnosis of renal parenchymal damage — This study is an observational study to evaluate the accuracy of renal parenchymal damage combined diagnosis with no intervention. All patients from the cohort accept MRI-DWI scan，the urinary biomarkers detection, disease gene detection and DMSA scan.
  1. This combined diagnosis includes MRI-DWI scan and the urinary biomarkers detection.
     MRI-DWI： All the scans are performed using the MagnetomVerio 3.0T magnetic resonance imaging system from Siemens.
     Urinary polypeptide collection: Urine samples requirements: volume between 50-100ml, specific gravity >1.010. Immunomagnetic beads isolation technique is used to collect polypeptide.
  2. The reference standard is DMSA scan: Intravenous injection of 99mTC-DMSA5mCi is followed by anterior and posterior planar imaging of the renal area 1 hour later. The DMSA scan images are read by 2 trained radiologists and confirmed by the special doctor of the center for diagnosis and treatment of renal and urinary diseases at the same time.

SUMMARY:
To establish the prediction of the renal damage and renal development deficiency in congenital anomalies of kidney and urinary tract (CAKUT), a diagnostic accuracy study on MRI-DWI combined with urinary microprotein detection is to carried out comparing with DMSA scan as the golden standard for renal damage.

DETAILED DESCRIPTION:
Congenital anomalies of kidney and urinary tract (CAKUT) is one of the common birth defects, with a morbidity of 6‰. The delayed diagnosis, due to its demanding diagnostic technique, may leads to long-term severe renal damage. This project is a prospective, continuous double-blind designed diagnostic accuracy study. The clinical diagnosis of CAKUT relies on a panel of radiological examinations most of which are invasive and risk of radiation harm for children. To establish the non-invasive and safe diagnosis detections of renal damage of CAKUT in children, a combination of MRI/DWI with urinary detection through Immunomagnetic beads isolation technique is to carried out to evaluate the renal deficiency in CAKUT comparing the dimercaptosuccinic acid (DMSA) scan as the golden standard of renal parenchymal damage. Analysis of sensitivity and specificity is to evaluate the accuracy of the combined diagnostic protocol. Furthermore the clinical information of pregnancy and phenotypes of the patients with CAKUT is to be collected with all the genetic information constructing the full phenotype- genotype spectrum for big data analysis and predictive model for early detection of renal damage in CAKUT.

ELIGIBILITY:
Inclusion Criteria:

Patient that was diagnosed clinically and genetically as:

* Renal parenchymal aplasia or ectopia, including simple renal aplasia,Multicystic Dysplastic Kidney, kidney tubules dysplasia, and hereditary cystic kidney. ①disease renal agenesis (RA): With ultrasound diagnosis of unilateral renal absence.②Renal hypoplasia (RH)/renal dysplasia (RD) is usually defined as renal volume less than two standard deviations of the average of the same age, or renal total volume less than 50% of the normal value of the same age. RD refers to the presence of undifferentiated or not metaplastic tissue in the kidney, with or without renal volume reduction. Diagnosis is based on the ultrasonic findings of multicystic dysplastic kidney (MCDK) and the diagnosis of unilateral or bilateral renal functional defects by means of isotopic renal functional imaging (DMSA or DTPA);
* Kidney tubular dysplasia: ①the diagnosis of polycystic kidney disease(ADPKD/ARPKD) is mainly dependent on imaging; Patients with a family history of ADPKD can be diagnosed with more than 3 renal cysts on either side. those who with bilateral renal diffuse enlargement with multiple cysts should be clinically considered with PKD even without family history of ADPKD, and relevant gene screening is recommended.②Simple renal cyst: single renal cyst was found by ultrasound or other imaging examination;③Nephronophthisis, NPHP: ultrasonography showed enhanced renal echo or unclear boundary between cortex and medulla, with or without genetic diagnosis or involvement of other system, gene sequence should be considered. Genetic molecular diagnosis is the main diagnostic basis of NPHP diagnosis.④nephrocalcinosis and urinary calculi: the diagnosis depends on the ultrasound diagnosis and the examinations of serum and urine electrolyte and metabolite should be performed to further diagnose the primary disease.
* Abnormalities of Ureter， renal pelvis and/or bladder: ① Dual collection system: Reduplication of kidney or renal pelvis/ureter depends on ultrasound, magnetic resonance imaging (MRI) diagnosis. ② Urinary obstruction: Including ureteropelvic junction obstruction, ureterovesical junction obstruction or insufficiency. The diagnosis of obstruction depends on magnetic resonance urography (MRU) and isotopic dynamic renal imaging(DTPA) ③ vesicoureteral reflux: The diagnosis depends on voiding cysternography (VCUG).
* Urinary tract anomalies: ① Urethral absence/urethra atresia/ectopic orifice: Diagnosis depends on physical examination and VCUG examination. ② Posterior urethral valve: Severe hydronephrosis can be found by ultrasound, and the diagnosis depends on VCUG examination.

Exclusion Criteria:

* Patient with renal failure due to different causes but without urine specimen;
* Other conditions that the researcher considers not suitable for inclusion

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric children diagnosed of CAKUT from Shanghai peri-conceptional parent-offspring cohort (SPCC) clinic research related outpatient and high-risk newborns referral outpatient, and those who are enrolled in nephrology department and urinary surgery department with CAKUT diagnosis.
Sampling Method: Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
The accuracy of combined diagnosis in evaluating renal parenchymal damage of CAKUT patients | Within 3 months since diagnosis of CAKUT.
  The accuracy of combined diagnosis includes sensitivity and specificity. The reference standard test (DMSA scan) and combined diagnosis are conducted in the cohort of pediatric children diagnosed of CAKUT.
  Sensitivity is defined as: The proportion of renal parenchymal damage is successfully screened out by combined diagnosis.
  Specificity is defined as: The proportion of children without renal parenchymal damage who are not recognized as impairment by combined diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China